CLINICAL TRIAL: NCT05967208
Title: Confidential Social Network Referrals for HIV Testing
Acronym: CONSORT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Duke University (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Principal Investigator, Jan Ostermann, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00120208
Record Dates: First submitted 2023-01-26; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONSORT referrals + Card referrals (Experimental): Intervention arm
  Interventions: Behavioral: CONSORT referrals; Behavioral: Card referrals
- Card referrals alone (Active Comparator): Control arm
  Interventions: Behavioral: Card referrals

INTERVENTIONS:
Behavioral: CONSORT referrals — Participants will be offered SMS-based confidential social network referrals for HIV testing ("CONSORT referrals") to extend to any of their social and sexual network contacts.
  Arms: CONSORT referrals + Card referrals
Behavioral: Card referrals — Participants will be offered physical invitation cards ("card referrals") to extend to any of their social and sexual network contacts.

SUMMARY:
Despite worldwide efforts to promote HIV testing, rates of testing remain low. The purpose of this study is to evaluate the acceptability, efficacy, and cost-effectiveness of confidential SMS-based social network referrals for HIV testing as a means of reaching high-risk individuals and prompting them to test for HIV. To accomplish this purpose, the study has 5 specific aims:

Aim 1 will conduct qualitative, formative work to identify desirable provider- and client-side characteristics of a confidential SMS-based HIV testing referral system.

Aim 2 will adapt an existing mHealth system (mParis) to add CONSORT functionality.

Aim 3 will pilot-test the CONSORT system to collect preliminary data on the system's acceptability, performance, and potential efficacy.

Aim 4 will evaluate the acceptability and efficacy of CONSORT in a randomized controlled trial.

Aim 5 will evaluate the incremental cost-effectiveness of CONSORT vs. other referral options.

If CONSORT is shown to be acceptable, effective, and cost-effective, such mobile-phone supported, chain-referral methods could greatly improve the cost-effectiveness of HIV testing efforts.

DETAILED DESCRIPTION:
No additional detail available

ELIGIBILITY:
Inclusion criteria:

* at least 18 years old
* live, work, or regularly receive care in Moshi, Tanzania
* literate

Exclusion criteria:

* under age 18 years
* does not live, work, or regularly receive care in Moshi, Tanzania
* illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of HIV testing | Within 30 days of the time of the testing offer
  The number of referred clients presenting for HIV testing at participating study sites within 30 days of the testing offer, per 100 index clients.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ostermann, PhD, Principal Investigator — University of South Carolina; Nathan Thielman, MD, Principal Investigator — Duke University; Bernard Njau, PhD, Principal Investigator — Kilimanjaro Christian Medical Centre, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
All investigators are committed to managing and distributing original data and results to enable subsequent availability to the scientific community, policy makers, and other stakeholders. Final research data including metadata and descriptors may be made available after publication of study findings through a CONSORT data repository. Researchers may access data by request to the Principal Investigators. Access will be provided subject to Tanzanian and US rules, laws, regulations and policies and consistent with institutional review board approvals and consent documents. If conditions prevent making some data elements available (e.g., third party data), relevant publications and presentations will be provided.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of study findings
Access Criteria: Access will be provided subject to Tanzanian and US rules, laws, regulations and policies and consistent with institutional review board approvals and consent documents. If conditions prevent making some data elements available (e.g., third party data), relevant publications and presentations will be provided.

REFERENCES:
- [Background] Ostermann J, Njau B, Masaki M, Mtuy T, Itemba D, Hobbie A, Yelverton V, Moore S, Yamanis T, Thielman NM. Feasibility, Acceptability, and Potential Cost-Effectiveness of a Novel Mobile Phone Intervention to Promote Human Immunodeficiency Virus Testing Within Social Networks in Tanzania. Sex Transm Dis. 2022 Nov 1;49(11):778-781. doi: 10.1097/OLQ.0000000000001611. Epub 2022 Jan 29. PMID 35093981
- [Derived] Ostermann J, Njau B, van Zwetselaar M, Yamanis T, McClimans L, Mwangi R, Beti M, Hobbie A, Gass SJ, Mtuy T, Thielman N. Mobile Phone-Based Confidential Social Network Referrals for HIV Testing (CONSORT): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 May 30;13:e55068. doi: 10.2196/55068. PMID 38814692